CLINICAL TRIAL: NCT01719341
Title: Study of Non-Myeloablative Haplo-identical Haematopoietic Stem Cell Transplantation in Patients With Haematological Malignancies or Acquired Aplastic Anaemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/00465
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Haematological Malignancies; Acquired Aplastic Anaemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Allogeneic haematopoietic stem cell transplantation (HSCT) is a potentially curative therapy for patients with both haematological and some non-haematological disorders. However, one of the major limiting factors for transplantation is the inability to identify a suitable HLA-matched donor. Development of an cost-effective and clinically efficacious alternative to HLA-identical sibling or unrelated donor transplantation would significantly expand the availability of allogeneic HSCT to patients in Singapore. Preliminary results indicate that the use of high dose post-transplant cyclophosphamide (Cy) for graft versus host disease (GVHD) prophylaxis in haplo-identical allogeneic HSCT is associated a low incidence of GVHD and low treatment related toxicity. We propose a phase II clinical trial to assess the efficacy of a haplo-identical allogeneic transplantation protocol using high dose post-transplant Cy for the treatment of patients with haematological disorders. A non-myeloablative protocol (Fludarabine-low dose cyclophosphamide-TBI) will be used for patients with bone marrow failure syndromes and indolent lymphoid disease. In view of the higher relapse risk of patients with myeloid malignancies, these patients will be treated with a reduced intensity conditioning regimen (Fludarabine-Busulphan). The primary end-point of the study will be overall survival at one year. Economic cost of the haplo-identical transplantation, as well as treatment timelines will be recorded and compared will other forms of unrelated donor allogeneic transplantation (umbilical cord blood transplantation and unrelated HLA-matched adult donor). Immunological reconstitution of patients following haplo-transplantation will be analysed and data will be utilized to guide future immunotherapy strategies post-transplantation.

One year survival after non-myeloablative haploidentical stem cell transplantation is not inferior to that observed after non-myeloablative volunteer unrelated donor or unrelated cord blood haematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

Patient Selection Inclusion criteria

1. Age under 70 years and older than 18 years
2. Absence of HLA fully compatible related donor
3. Need for an urgent transplantation, defined as within 8 weeks of referral to the transplant centre or absence of HLA-compatible VUD after searching the international registries. Patients with a HLA-compatible VUD but whose donor is considered by the transplantation centre as unsuitable will also be eligible. 4. Informed consent.

Disease inclusion criteria:

In general this encompasses all haematological disorders where a volunteer unrelated donor (UD) transplant is clinically indicated.

1. Acute, chronic leukaemia or myelodysplastic syndrome for which allogeneic transplantation is considered as the best treatment option.

a. Acute myeloid leukaemia (AML) i. In first complete remission (CR1) with one of the following characteristics:

1. High risk cytogenetic or molecular alterations (e.g. t(9;22), deletion 7/7q-, monosomy 5 or del(5q), 3q26 alterations, complex karyotype [3 or more anomalies], p53 alterations, 11q23 especially t(6;11) abnormalities, FLT-3 ITD, monosomal karyotype.
2. Leukocytes at diagnosis > 50 x109/l (except in cases with good prognosis molecular rearrangements for which leukocytes should be > 100 x 109/l) b. Myelodysplastic syndromes1. International Prognosis Index (IPSS) above 1 (intermediate group 2 or high risk)

2. IPSS 0 or 0.5 in the presence of cytopenias requiring treatment. c. Therapy related AML or MDS in first CRd. AML or MDS in second (CR2) or subsequent CRe. Ph'-positive chronic myeloid leukaemia i. In first chronic phase if refractory and/or intolerance to tyrosine kinase inhibitors is clearly demonstrated ii. In second chronic phase 2. Acute lymphoblastic leukaemia (ALL)a. In CR1 with one of the following characteristics: i. Very high risk chromosome or molecular alterations (e.g. t(9;22), t(4;11), complex karyotype in adults, bcr/abl rearrangements, MLL rearrangements) ii. Slow response to induction treatment defined as the presence of >10% blasts in bone marrow at day 14 of induction treatmentiii. Adults aged > 30 yearsiv. Adults with B ALL cell line with a number of leukocytes at diagnosis >25 x 109/L or T ALL cell line with a number of leukocytes at diagnosis >100X109/Lb. In CR2 or subsequent CR 3. Non-Hodgkin's lymphomaa. Follicular NHL: in second or subsequent complete or partial remissionb. Mantle cell NHL: in second or subsequent complete or partial remissionc. High grade NHL: in second complete or very good partial remission 4. Hodgkin's diseasea. in second or subsequent complete or partial remission 5. Chronic lymphocytic leukaemia. a. in second or subsequent remissionb. with adverse risk prognostic features in first remission 6. Acquired Aplastic Anaemia 7. Myelofibrosis- Lille score -high, Cervantes score-high 8. Other haematological malignancies for which UD HSCT is indicated

Exclusion Criteria:

1. Patients with an available 7-8/8 HLA-A, -B, -C, -DRB1 matched sibling donor or 7-8/8 unrelated bone marrow donor
2. Availability of suitable UCB unit/s and eligible for an UCB transplant
3. ECOG performance status worse than 2
4. Cardiac insufficiency requiring treatment, symptomatic coronary artery disease or LVEF less than 35%.
5. Hepatic disease, with total bilirubin greater than 2 times upper limit of normal or AST > 5 times upper limit of normal.
6. Severe hypoxaemia, pO2 < 70 mm Hg, with decreased DLCO < 50% of predicted; or mild hypoxemia, pO2 < 80 mm Hg with severely decreased DLCO < 50% of predicted.
7. Impaired renal function (creatinine > 2 times upper limit of normal or creatinine clearance < 50% for age, gender, weight).
8. Previous irradiation that precludes the safe administration of an additional dose of 200 cGy of total body irradiation (TBI).
9. HIV positive patients.
10. Female patients who are pregnant or breast feeding due to risks to foetus from conditioning regimen and potential risks to nursing infants.
11. Life expectancy severely limited by diseases other than the disease indication for transplant
12. Serious concurrent uncontrolled infection e.g. active tuberculosis, mycoses or viral infection
13. Serious psychiatric/ psychological disorders
14. Absence of /inability to provide informed consent
15. Patients with acute leukaemia with >5% bone marrow blasts
16. Intermediate or high grade NHL, mantle cell NHL and Hodgkin's disease that is refractory to salvage therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample size estimation based on Case and Morgan Two Stage Phase II Design with an expected duration of accrual of 2 years, assuming a power of 80% and a level of significance of 10%. With an S0 of 0.25 and SA of 0.50, an interim analysis will be performed after 14 patients are recruited with an anticipated final recruitment total of 21 patients for each arm of the study.
Sampling Method: Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
1 year overall survival after HLA-Haploidentical transplantation | 1 year

SECONDARY OUTCOMES:
Progression free survival one and 2 years post-transplantation | 2 years
Cumulative incidence of relapse/progression at one and 2 years post-transplant | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Zi Yi Lim, MB ChB, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Aversa F. Haploidentical haematopoietic stem cell transplantation for acute leukaemia in adults: experience in Europe and the United States. Bone Marrow Transplant. 2008 Mar;41(5):473-81. doi: 10.1038/sj.bmt.1705966. Epub 2008 Jan 7. PMID 18176612
- [Background] Luznik L, Bolanos-Meade J, Zahurak M, Chen AR, Smith BD, Brodsky R, Huff CA, Borrello I, Matsui W, Powell JD, Kasamon Y, Goodman SN, Hess A, Levitsky HI, Ambinder RF, Jones RJ, Fuchs EJ. High-dose cyclophosphamide as single-agent, short-course prophylaxis of graft-versus-host disease. Blood. 2010 Apr 22;115(16):3224-30. doi: 10.1182/blood-2009-11-251595. Epub 2010 Feb 2. PMID 20124511